CLINICAL TRIAL: NCT04509635
Title: A Single-centre, Prospective, Randomised, Controlled, Unblinded, Parallel-group Trial of Cetuximab Plus Chemotherapy Versus Chemotherapy Alone for Colorectal Cancer Liver Metastasis With Progression After First-line Treatment of Cetuximab
Brief Title: Cetuximab Re-challenge for Colorectal Cancer Liver Metastasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cet-rechallenge
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Liver Metastases; Cetuximab
Keywords: Colorectal Cancer; Liver Metastases; Cetuximab; Re-challenge
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Using treatment of cetuximab plus chemotherapy. Cetuximab: 500 mg/m2 IV over 2 hours, day 1, every 2 weeks. Chemotherapy: detailed regimen is determined by a multi-disciplinary team.
  Interventions: Drug: Cetuximab; Drug: Chemotherapy
- Arm B (Active Comparator): Using treatment of chemotherapy alone. Chemotherapy: detailed regimen is determined by a multi-disciplinary team
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Cetuximab — Cetuximab is used for only patients with ctDNA test RAS wild type.
  Arms: Arm A
Drug: Chemotherapy — The detailed regimen is determined by a multi-disciplinary team according to the previous use of chemotherapy.

SUMMARY:
For patients with unresectable colorectal cancer liver metastases, preclinical studies have shown that after the resistance of cetuximab, the treatment sensitivity can be restored by stopping cetuximab for a period of time. This is called the cetuximab re-challenge. And the circulating tumor DNA (ctDNA) test is reported a biomarker for the efficacy of cetuximab rechallenge. However, there is still no randomized controlled trial for verification. This study aims at patients after the first-line treatment of cetuximab has progressed. After the second-line non-cetuximab treatment has progressed, the effects of re-application of combined with cetuximab and chemotherapy alone are compared to verify the re-challenge effect.

DETAILED DESCRIPTION:
Patients with colorectal cancer liver metastases were RAS wild type, received first-line cetuximab plus chemotherapy. After first-line progression, second-line non-cetuximab treatment were used. After second-line progression, ctDNA is test, and patients with RAS wild-type are enrolled in the study to compare cetuximab plus chemotherapy vs. chemotherapy alone as third-line treatment. Treatment will continue until disease progression or unacceptable toxic effects. The primary endpoint is the disease control rate，which will be assessed by local multidisciplinary team with the use of contrast-enhanced CT or MRI after 4 cycles and then every other 4 cycles up to 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Primary tumour was histologically confirmed colorectal adenocarcinoma;
2. Clinical or radiological evidence of non-resectable liver metastases;
3. With at least one measurable tumor;
4. Received first-line cetuximab (RAS gene wild type) treatment and progressed
5. Received second-line non-cetuximab treatment and progressed
6. Received circulating tumor DNA test and has RAS gene wild type status;
7. Performance status (ECOG) 0~1
8. A life expectancy of ≥ 3 months
9. Adequate hematological function: Neutrophils≥1.5 x109/l and platelet count≥100 x109/l; Hb ≥9g/dl (within 1 week prior to randomization)
10. Adequate hepatic and renal function: Serum bilirubin≤1.5 x upper limit of normal (ULN), alkaline phosphatase ≤5x ULN, and serum transaminase (either aspartate transaminase (AST) or alanine transaminase (ALT)) ≤ 5 x ULN(within 1 week prior to randomization);
11. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Patients with known hypersensitivity reactions to any of the components of the study treatments.
2. Acute or sub-acute intestinal occlusion
3. Pregnancy (absence confirmed by serum/urine β-HCG) or breast-feeding
4. Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix Known drug abuse/ alcohol abuse
5. Legal incapacity or limited legal capacity
6. Pre-existing peripheral neuropathy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
disease control rate | 2 years
  According to the RECIST v.1.1, the disease control rate (DCR) is the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD), evaluated by radiology (CT, MRI, etc.).

SECONDARY OUTCOMES:
objective response rate | 2 years
  According to the RECIST v.1.1, the disease control rate (DCR) is the proportion of patients with complete response (CR) and partial response (PR), evaluated by radiology (CT, MRI, etc.).
progression-free survival | 2 years
  The period from the first day of treatment to the date of disease progression (PD) or to death.
overall survival | 2 years
  The period from the first day of treatment to the date of death.

IPD SHARING:
Plan to Share IPD: Undecided